CLINICAL TRIAL: NCT03640455
Title: Etude Pilote Randomisee Versus Placebo Evaluant l'Efficacite de la Stimulation Electrique Transcranienne de Faible Intensite (Tdcs) Dans le Soulagement de la Dyspnee Chez Les Patients Sous Ventilation Mecanique en Reanimation
Brief Title: Randomized Study Evaluating the Efficacy of Low Intensity Transcranial Electrical Stimulation (Tdcs) for the Relief of Dyspnea
Acronym: tDCS-DYSP-REA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K160904
Record Dates: First submitted 2018-07-09; First posted 2018-08-21 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Dyspnea; Mechanical Ventilation Complication
MeSH Terms: conditions — Dyspnea | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): A tDCS (Low Current Transcranial Stimulation) device with two electrodes: active and reference, will be used. The tDCS will be applied next to the cortical representation zone of the primary motor cortex and left pre-motor for 30 minutes; dummy stimulation will be given.
  Interventions: Device: Placebo
- Anodal tDCS (Experimental): A tDCS (Low Current Transcranial Stimulation) device with two electrodes: active and reference, will be used. The tDCS will be applied next to the cortical representation zone of the primary motor cortex and left pre-motor for 30 minutes; Current Transcranial Stimulation (intensity 2 mA) will be given in anodal polarity.
  Interventions: Device: Anodal
- Cathodal tDCS (Experimental): A tDCS (Low Current Transcranial Stimulation) device with two electrodes: active and reference, will be used. The tDCS will be applied next to the cortical representation zone of the primary motor cortex and left pre-motor for 30 minutes; Current Transcranial Stimulation (intensity 2 mA) will be given in cathodal polarity.
  Interventions: Device: Cathodal

INTERVENTIONS:
Device: Placebo — A tDCS (Low Current Transcranial Stimulation) device with two electrodes: active and reference, will be used. The tDCS will be applied next to the cortical representation zone of the primary motor cortex and left pre-motor for 30 minutes; placebo (dummy stimulation), according to the patient's randomization arm.
  Arms: Placebo
Device: Anodal — A tDCS (Low Current Transcranial Stimulation) device with two electrodes: active and reference, will be used. The tDCS will be applied next to the cortical representation zone of the primary motor cortex and left pre-motor for 30 minutes; intensity 2 mA, in anodal polarity, according to the patient's randomization arm.
  Arms: Anodal tDCS
Device: Cathodal — A tDCS (Low Current Transcranial Stimulation) device with two electrodes: active and reference, will be used. The tDCS will be applied next to the cortical representation zone of the primary motor cortex and left pre-motor for 30 minutes; intensity 2 mA, in cathodal polarity, according to the patient's randomization arm.
  Arms: Cathodal tDCS

SUMMARY:
Nearly half (47%) of patients with mechanical ventilation in the intensive care unit report having dyspnea. This respiratory distress, with a feeling of "thirst for air", often reaches unbearable limits and is a major factor in the deterioration of the quality of life and the prognosis of patients. Physiopathological mechanisms of dyspnea are beginning better understood and have analogies with those of pain. Like pain, dyspnea often persists despite appropriate treatment of the cause, because of perceptual dysfunction related to changes in cortical excitability and neuronal plasticity and requires specific treatments. Studies have shown that Transcranial Stimulation by low Current (tDCS) was able to modulate the perception of acute pain induced and chronic pain. The tDCS modulates the functioning of a whole set of brain structures including the anterior cingulate gyrus, the prefrontal cortex, the thalamus and the brain stem, some of which have an established role in the central integration of pain and dyspnea. The investigators have recently demonstrated that the application of tDCS on the primary cortical motor area reduces the excitability of the central neurological pathways dedicated to the respiratory muscles in healthy subjects. The investigators therefore hypothesize that tDCS could relieve dyspnea in intensive care. In this research project, the investigators propose to evaluate the efficiency of tDCS on dyspnea in patients admitted to intensive care unit, having sepsis and mechanically ventilated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, hospitalized in intensive care unit, presenting a sepsis, having required a mechanical ventilation since at least 24h.
* Non-sedated or showing good wake up (Richmond Agitation-Sedation Scale score (RASS)> -3 at inclusion (Sessler et al., 2002)) within 48 hours after cessation of sedation
* Patient able to answer by "yes" or "no" to simple questions
* Showing significant dyspnea (level ≥ 4) on the A1 sub-scale of the Multidimensional Dyspnea Profile (MPD-A1 ≥ 4).
* Signature of informed consent by the patient or his relative.

Exclusion Criteria:

* Patient under guardianship,
* Wake up delay, coma (GCS ≤ 8), or severe agitation.
* chronic respiratory pathology
* respiratory pathology, neuromuscular or neuro-sensory disability (auditory or visual).
* Cranioplasty
* Language barrier, refusal to participate in the study or to sign the informed consent,
* Pregnant or nursing woman,
* No affiliation to a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-05-09 (Actual); Study Completion 2022-01-09 (Estimated)

PRIMARY OUTCOMES:
Differential of the Dyspnea | 30 min
  Assessing differential of the Dyspnea Multidimensional Profile (MPD-A1) Scale A1 (from 0 to 10): between before (30 min before) and after (30 min after) the use of tDCS.
  The scale name is " Multidimensional dyspnea profile". The A1 dimension will be used and measures affective dimensions unpleasantness and overall breathing discomfort. The minimum score is 0 ( neutral) and the maximum score is 10 (unbearable discomfort).

SECONDARY OUTCOMES:
Differential of the QS | 30 min
  Assessing differentials of the QS of the Multidimensional Dyspnea Profile measured between before and after the tDCS (MPD-QS scales) between before (30 min before) and after (30 min after) the use of tDCS.
Differential of the A2 dimension | 30 min
  Assessing differentials of the sale A2 of the Multidimensional Dyspnea Profile measured between before and after the tDCS (MPD-A2 scales) between before (30 min before) and after (30 min after) the use of tDCS.
Differential of IC-RDOS | 30 min
  Differential of Diagnostic Accuracy of Respiratory Distress Observation Scales (IC-RDOS scale) between before (30 min before) and after (30 min after) the use of tDCS.
  Persichini, R., Gay, F., Schmidt, M., Mayaux, J., Demoule, A., Morélot-Panzini, C., & Similowski, T. (2015). Diagnostic accuracy of respiratory distress observation scales as surrogates of dyspnea self-report in intensive care unit patients. Anesthesiology: The Journal of the American Society of Anesthesiologists, 123(4), 830-837.
Pre-inspiratory potentials (PIP) | 1 day
  Presence of possible PIP on Electroencephalography (EEG)
Death | 28 days
Delirium | 28 days
  Cumulative incidence of delirium and its duration
Mechanical ventilation | 28 days
  Cumulative incidence of mechanical ventilation
ICU length of stay | 28 days

OTHER OUTCOMES:
mouth pressure | 30 min
  differences of mouth pressure between before (30 min before) and after (30 min after) the use of tDCS
respiratory rate | 30 min
  differences of respiratory rate between before (30 min before) and after (30 min after) the use of tDCS
tidal volume | 30 min
  differences of tidal volume between before (30 min before) and after (30 min after) the use of tDCS

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Raymond Poincaré, Garches, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Azabou E, Bao G, Heming N, Bounab R, Moine P, Chevallier S, Chevret S, Resche-Rigon M, Siami S, Sharshar T, Lofaso F, Annane D. Randomized Controlled Study Evaluating Efficiency of Low Intensity Transcranial Direct Current Stimulation (tDCS) for Dyspnea Relief in Mechanically Ventilated COVID-19 Patients in ICU: The tDCS-DYSP-COVID Protocol. Front Med (Lausanne). 2020 Jun 26;7:372. doi: 10.3389/fmed.2020.00372. eCollection 2020. PMID 32671084